CLINICAL TRIAL: NCT06473064
Title: Evaluation of Feasibility and Aesthetic Outcomes of Benelli Technique for Nipple Sparing Mastectomy in Surgical Treatment of Grade 3 and 4 Gynecomastia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ezzat Essam Ezzat Osman, resident at general surgery department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Benelli technique gynecomastia
Record Dates: First submitted 2024-05-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Surgical Managment of Gynecomastia
MeSH Terms: interventions — Mastectomy, Subcutaneous

STUDY DESIGN:
Intervention Model Description: * The Nipple areola complex (NAC )margins on both sides are marked as circular.
    * Around the initial circle, a second circle (external) was drawn 1 cm broader than the boundary.
    * The skin was resected, with deepithelialization between the two circles.
    * A transdermal incision was made through the border of the external circle.
  * The breast tissue around the pedicle was lifted over the pectoral fascia and excised by preserving the NAC and the underlying breast pedicle
    -The base of the mammary pedicle under the NAC was infixed at the farthest end of the mastectomy area by using 3/0 absorbable multifilament suture material
  * Hence, the space formed after mastectomy was filled with a breast pedicle located posterior to the NAC.
  * The closure of the circular deepithelialized area around the NAC with a diameter of 1 cm accomplished by using 4/0 absorbable monofilament suture material and the surgery was completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- grade 3 and 4 gynecomastia (Other): To evaluate and determine the posibility of complication of benelli technique for nipple sparing mastectomy in surgical treatment of grade 3and 4 gynecomastia and its cosmetic effect
  Interventions: Other: Benelli technique for nipple sparing mastectomy in surgical treatment of grade 3 and 4 gynecomastia

INTERVENTIONS:
Other: Benelli technique for nipple sparing mastectomy in surgical treatment of grade 3 and 4 gynecomastia — .The Nipple areola complex (NAC )margins on both sides are marked as circular. -Around the initial circle, a second circle (external) was drawn 1 cm broader than the boundary.
  * The skin was resected, with deepithelialization between the two circles.
  * A transdermal incision was made through the border of the external circle.
    -. The breast tissue around the pedicle was lifted over the pectoral fascia and excised by preserving the NAC and the underlying breast pedicle
  * The base of the mammary pedicle under the NAC was infixed at the farthest end of the mastectomy area by using 3/0 absorbable multifilament suture material
    * Hence, the space formed after mastectomy was filled with a breast pedicle located posterior to the NAC.
    * The closure of the circular deepithelialized area around the NAC with a diameter of 1 cm accomplished by using 4/0 absorbable monofilament suture material and the surgery was completed

SUMMARY:
Gynecomastia is the benign proliferation of male breast tissue caused by an increase in the estrogen/androgen activity ratio. It manifests itself physiologically (adolescence, puberty, and old age) as well as pathologically (androgen insufficiency caused by drugs or disease, testicular tumors, hyperthyroidism, and chronic renal failure).

* In spite of the variety of methods and tools such as (liposuction and circumareolar inframammary inscion ) used in gynecomastia surgery, in gynecomastia the results are satisfactory in grades 1 and 2 while grades 3 and 4 gynecomastia present a surgical challenge.
* As some postoperative frustrating problems still cannot be completely eliminated, the most common of these are a saucer-like deformity (over resection under areola), bleeding, followed by seroma, infection, ischemic necrosis of nipple areola complex residual gynecomastia (under resection), persistence of inframammary fold, contour irregularities, and asymmetries between breasts.
* the objective, in this research, is to demonstrate the The role of Benelli technique in removal of gynecomastia grade 3 and grade 4 in clinical and cosmetic outcomes

DETAILED DESCRIPTION:
• The aim of this study the investigator determines the feasibility and cosmetic outcomes of Benelli technique for nipple sparing mastectomy in cases of grade 3 and 4 gynecomastia

ELIGIBILITY:
Inclusion Criteria:

* adult male complaining of unilateral or bilateral grade 3 and 4 gynecomastia
* pseudo gynecomastia following massive weight loss with excess skin and laxity

Exclusion Criteria:

* patients with chronic liver failure
* hyperthyroidism
* Malignant mass
* Diabetics
* smokers
* patients with medical treatment as anabolic steroids .

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-10-19 (Estimated)

PRIMARY OUTCOMES:
Benelli technique for nipple sparing mastectomy in surgical treatment of grade 3 and 4 gynecomastia | baseline
  to evaluate and determine the feasibility and complications of benelli techniques for nipple sparing mastectomy in surgical tratment of grade 3 and 4 gynecomastia and also its cosmetic effect

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Result] Benelli L. A new periareolar mammaplasty: the "round block" technique. Aesthetic Plast Surg. 1990 Spring;14(2):93-100. doi: 10.1007/BF01578332. PMID 2185619
- [Result] Tarallo M, Di Taranto G, Fallico N, Ribuffo D. The round-the-clock technique for correction of gynecomastia. Arch Plast Surg. 2019 May;46(3):221-227. doi: 10.5999/aps.2018.00472. Epub 2019 May 15. PMID 31113185
- [Result] Colombo-Benkmann M, Buse B, Stern J, Herfarth C. Indications for and results of surgical therapy for male gynecomastia. Am J Surg. 1999 Jul;178(1):60-3. doi: 10.1016/s0002-9610(99)00108-7. PMID 10456706
- [Result] Letterman G, Schurter M. Suggested nomenclature for aesthetic and reconstructive surgery of the breast. Part III: Gynecomastia. Aesthetic Plast Surg. 1986;10(1):55-7. doi: 10.1007/BF01575270. No abstract available. PMID 3087145